CLINICAL TRIAL: NCT00002318
Title: Randomized, Comparative Trial of DOX-SL (Stealth Liposomal Doxorubicin Hydrochloride) Versus Adriamycin, Bleomycin, and Vincristine (ABV) in the Treatment of Severe AIDS-Related Kaposi's Sarcoma
Brief Title: A Comparison of DOX-SL Versus Adriamycin Plus Bleomycin Plus Vincristine in the Treatment of Severe AIDS-Related Kaposi's Sarcoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sequus Pharmaceuticals (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Model: Parallel | Purpose: Treatment
Other Study IDs: 134A; LTI-30-10
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1996-01

CONDITIONS: Sarcoma, Kaposi; HIV Infections
Keywords: Vincristine; Sarcoma, Kaposi; Liposomes; Doxorubicin; Drug Therapy, Combination; Acquired Immunodeficiency Syndrome; Bleomycin; Drug Carriers
MeSH Terms: conditions — Sarcoma, Kaposi; HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Doxorubicin; Liposomes; Bleomycin; Vincristine

INTERVENTIONS:
Drug: Doxorubicin hydrochloride (liposomal)
Drug: Bleomycin sulfate
Drug: Vincristine sulfate
Drug: Doxorubicin hydrochloride

SUMMARY:
To determine the efficacy of Stealth liposomal doxorubicin hydrochloride (DOX-SL) in the treatment of severe AIDS-related Kaposi's sarcoma (KS) by comparison with the established therapy ABV: Adriamycin (doxorubicin)/bleomycin/vincristine. To evaluate the safety and tolerance of DOX-SL compared to ABV in a population of AIDS patients with severe KS.

DETAILED DESCRIPTION:
Patients are randomized to receive either DOX-SL or the ABV combination. Infusions are given on day 1 and every 2 weeks for a total of six cycles. Kaposi's sarcoma lesions are evaluated prior to every cycle, at the end of the last treatment cycle, and 4 weeks following the end of the last treatment. Patients must agree to have one or more representative KS lesions biopsied.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Prophylaxis for PCP, cryptococcal, and herpes infections, and antiretroviral therapy (e.g., AZT, ddC, ddI) provided these doses have been stable for at least 1 month.
* Therapy for tuberculosis, fungal, and herpes infections except with potentially myelotoxic chemotherapy.
* Foscarnet for new episodes of cytomegalovirus infection.
* Colony-stimulating factors and erythropoietin.

Patients must have:

* Biopsy-proven, progressive, AIDS-related Kaposi's sarcoma, with any of the following:
* At least 25 mucocutaneous lesions.
* Ten or more new lesions in the prior month.
* Documented visceral disease with at least two accessible cutaneous lesions.
* Two accessible cutaneous lesions with edema.
* Documented anti-HIV antibody.
* No active opportunistic infection with mycobacteria, cytomegalovirus, toxoplasma, Pneumocystis carinii, or other microorganisms (if under treatment with myelotoxic drugs).
* Life expectancy > 4 months.

NOTE:

* Patients who respond to therapy on this protocol, as well as those who fail the ABV combination, are eligible to enter the Liposome Technology open trial using DOX-SL alone.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Clinically significant cardiac, hepatic, or renal disease.
* Peripheral neuropathy, signs of moderate to severe sensory loss, or moderate to marked motor loss.
* Inability to comply with the study.

Concurrent Medication:

Excluded:

* Other cytotoxic chemotherapy.
* Ganciclovir.

Patients with the following prior conditions are excluded:

* Prior neoplasms treated with extensive chemotherapy that, in the investigator's opinion, has led to irreversibly compromised bone marrow function.
* History of idiosyncratic or allergic reaction to bleomycin or vincristine.

Prior Medication:

Excluded:

* Prior anthracycline therapy.
* Cytotoxic chemotherapy or interferon treatment within the past 4 weeks.

Prior Treatment:

Excluded:

* Radiation or electron beam therapy within the past 3 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225

CONTACTS AND LOCATIONS:
Locations (27):
- United States (27):
  - East Bay AIDS Ctr, Berkeley, California
  - Pacific Oaks Med Group, Beverly Hills, California
  - Hematology - Oncology Med Group of San Fernando Valley, Encino, California
  - Dr Becky Miller, Los Angeles, California
  - Apogee Med Group, San Diego, California
  - UCSF - San Francisco Gen Hosp, San Francisco, California
  - Kaiser Permanente Med Ctr, San Francisco, California
  - UCSF, San Francisco, California
  - San Francisco Veterans Administration Med Ctr, San Francisco, California
  - Pacific Oaks Med Group, Sherman Oaks, California
  - Dr Mahmoud Mustafa, Washington D.C., District of Columbia
  - Univ of Miami School of Medicine, Miami, Florida
  - H Lee Moffit Cancer Ctr and Research Institute, Tampa, Florida
  - American Med Research Institute, Atlanta, Georgia
  - Infectious Disease Rsch Consortium of GA / SE Clin Resources, Atlanta, Georgia
  - Northwestern Med Faculty Foundation, Chicago, Illinois
  - Rush Presbyterian Med College, Chicago, Illinois
  - Illinois Masonic Med Ctr / The Cancer Ctr, Chicago, Illinois
  - Henry Ford Hosp, Detroit, Michigan
  - Washington Univ, St Louis, Missouri
  - Roswell Park Cancer Institute, Buffalo, New York
  - Saint Vincent's Hosp and Med Ctr, New York, New York
  - New York Univ Med Ctr, New York, New York
  - Saint Luke's - Roosevelt Hosp Ctr, New York, New York
  - Graduate Hosp / Tuttleman Cancer Ctr, Philadelphia, Pennsylvania
  - Comprehensive Care Ctr, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas

REFERENCES:
- [Background] Gill PS, Wernz J, Scadden DT, Cohen P, Mukwaya GM, von Roenn JH, Jacobs M, Kempin S, Silverberg I, Gonzales G, Rarick MU, Myers AM, Shepherd F, Sawka C, Pike MC, Ross ME. Randomized phase III trial of liposomal daunorubicin versus doxorubicin, bleomycin, and vincristine in AIDS-related Kaposi's sarcoma. J Clin Oncol. 1996 Aug;14(8):2353-64. doi: 10.1200/JCO.1996.14.8.2353. PMID 8708728